CLINICAL TRIAL: NCT03740035
Title: Adaptation of an eHealth (Web-application) Platform for Delivery of a Sedentary Behavior Intervention Among Prostate Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Pl left institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00051239; CCCWFU 04118 (Other: NCI); P30CA012197 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Sedentary Lifestyle
Keywords: Prostate Cancer; eHealth; movement
MeSH Terms: conditions — Sedentary Behavior; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Prostate cancer patients that who have been actively receiving care through Wake Forest Baptist Comprehensive Cancer Center and/or satellite clinics over the past two-year period will be using an eHealth for Sedentary Behavior.
  Interventions: Device: eHealth for Sedentary Behavior

INTERVENTIONS:
Device: eHealth for Sedentary Behavior — Prostate cancer patients will be testing the usability and acceptability of the eHealth web app for sedentary behavior

SUMMARY:
The overall objective of this study is to adapt and refine an existing eHealth (web-application/web-app/app) platform designed to promote spontaneous movement (reducing sedentary behavior) among older adults, to men with prostate cancer.

DETAILED DESCRIPTION:
Primary treatments for prostate cancer (PCa) accelerate aging-related changes in body composition and declines in physical function and quality of life ; the median age at PCa diagnosis is 66 years and approximately 64% of PCa survivors are > 70 years. The negative side effects of treatments are pronounced in older, sedentary, overweight or obese men with existing comorbidities. The concomitant loss of skeletal muscle mass, increased deposition of adipose tissue and loss of bone mineral density leads to fractures, cancer-related fatigue, frailty, compromised physical functioning, disability and loss of independence as well as anxiety and depression. Regular physical activity reduces morbidity, improves survival and can buffer PCa patients against the negative side-effects of treatment, yet less than 20% are meeting recommended guidelines-and most spend up to 70% of their time each day in sedentary behavior. Targeting a reduction in sedentary behavior by promoting regular spontaneous movement in conjunction with regular resistance training may be an effective approach for PCa patients who are likely to be fatigued and functionally impaired. Traditional theory-based exercise interventions have shown preliminary efficacy for promoting short-term exercise, but can be improved for longer-term efficacy. Traditional exercise interventions are generally not individually tailored, and therefore cannot incorporate behavioral theory to re-engage participants when lapses in self-regulation occur. eHealth technologies can enhance traditional theory-based exercise interventions. The study team hypothesizes that an eHealth delivered intervention can effectively facilitate the development and maintenance of self-regulatory skills that are critical to sustaining long-term behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer.
* Currently (in last 2-years) receiving care for prostate cancer at WFBMC.
* Currently owns a smartphone or a tablet computer (iOS and major brand Android devices not including eReaders).
* English-speaking.

Exclusion Criteria:

* Unable to provide informed consent (e.g., delirium).
* Unable to ambulate safely (fall risk).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men with biological male reproductive organs
Study Population: Prostate cancer patients currently receiving treatment
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Assessment of the design features and functionality of the web-app | 45 minutes
  Participants will be given qualitative interviews on the functionality of the web-app. A thematic content analysis (TCA) for the evaluation of Think-Aloud and interview data will be used. Transcripts will be imported into ATLAS.ti software (Version 8, Berlin, Germany) and reviewed by the study team using an iterative approach.
System Usability Scale | 30 minutes
  Participants will answer 10, 5-point Likert-type questions to collect perceptions of the usability of the web-app. Total score 10-50, Higher scores denote better outcomes
Participant reflection on web-app features | 30 minutes
  Descriptive statistics to report on the open-ended qualitative reflections on app features will be coded using thematic content anaylsis as audio recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda L Bitting, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Chambers SK, Ng SK, Baade P, Aitken JF, Hyde MK, Wittert G, Frydenberg M, Dunn J. Trajectories of quality of life, life satisfaction, and psychological adjustment after prostate cancer. Psychooncology. 2017 Oct;26(10):1576-1585. doi: 10.1002/pon.4342. Epub 2017 Jan 11. PMID 27943512
- [Background] Cheung AS, Zajac JD, Grossmann M. Muscle and bone effects of androgen deprivation therapy: current and emerging therapies. Endocr Relat Cancer. 2014 Oct;21(5):R371-94. doi: 10.1530/ERC-14-0172. Epub 2014 Jul 23. PMID 25056176
- [Background] Alibhai SM, Duong-Hua M, Cheung AM, Sutradhar R, Warde P, Fleshner NE, Paszat L. Fracture types and risk factors in men with prostate cancer on androgen deprivation therapy: a matched cohort study of 19,079 men. J Urol. 2010 Sep;184(3):918-23. doi: 10.1016/j.juro.2010.04.068. PMID 20643458
- [Background] Pirl WF, Greer JA, Goode M, Smith MR. Prospective study of depression and fatigue in men with advanced prostate cancer receiving hormone therapy. Psychooncology. 2008 Feb;17(2):148-53. doi: 10.1002/pon.1206. PMID 17443645
- [Background] Bylow K, Dale W, Mustian K, Stadler WM, Rodin M, Hall W, Lachs M, Mohile SG. Falls and physical performance deficits in older patients with prostate cancer undergoing androgen deprivation therapy. Urology. 2008 Aug;72(2):422-7. doi: 10.1016/j.urology.2008.03.032. Epub 2008 Jun 17. PMID 18561991
- [Background] Dinh KT, Reznor G, Muralidhar V, Mahal BA, Nezolosky MD, Choueiri TK, Hoffman KE, Hu JC, Sweeney CJ, Trinh QD, Nguyen PL. Association of Androgen Deprivation Therapy With Depression in Localized Prostate Cancer. J Clin Oncol. 2016 Jun 1;34(16):1905-12. doi: 10.1200/JCO.2015.64.1969. Epub 2016 Apr 11. PMID 27069075
- [Background] Bhatia N, Santos M, Jones LW, Beckman JA, Penson DF, Morgans AK, Moslehi J. Cardiovascular Effects of Androgen Deprivation Therapy for the Treatment of Prostate Cancer: ABCDE Steps to Reduce Cardiovascular Disease in Patients With Prostate Cancer. Circulation. 2016 Feb 2;133(5):537-41. doi: 10.1161/CIRCULATIONAHA.115.012519. No abstract available. PMID 26831435
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Richman EL, Kenfield SA, Stampfer MJ, Paciorek A, Carroll PR, Chan JM. Physical activity after diagnosis and risk of prostate cancer progression: data from the cancer of the prostate strategic urologic research endeavor. Cancer Res. 2011 Jun 1;71(11):3889-95. doi: 10.1158/0008-5472.CAN-10-3932. Epub 2011 May 24. PMID 21610110
- [Background] Kenfield SA, Stampfer MJ, Giovannucci E, Chan JM. Physical activity and survival after prostate cancer diagnosis in the health professionals follow-up study. J Clin Oncol. 2011 Feb 20;29(6):726-32. doi: 10.1200/JCO.2010.31.5226. Epub 2011 Jan 4. PMID 21205749
- [Background] Thorsen L, Courneya KS, Stevinson C, Fossa SD. A systematic review of physical activity in prostate cancer survivors: outcomes, prevalence, and determinants. Support Care Cancer. 2008 Sep;16(9):987-97. doi: 10.1007/s00520-008-0411-7. Epub 2008 Feb 15. PMID 18274783
- [Background] Galvao DA, Newton RU, Gardiner RA, Girgis A, Lepore SJ, Stiller A, Occhipinti S, Chambers SK. Compliance to exercise-oncology guidelines in prostate cancer survivors and associations with psychological distress, unmet supportive care needs, and quality of life. Psychooncology. 2015 Oct;24(10):1241-1249. doi: 10.1002/pon.3882. Epub 2015 Jun 18. PMID 26087455
- [Background] Blanchard CM, Courneya KS, Stein K; American Cancer Society's SCS-II. Cancer survivors' adherence to lifestyle behavior recommendations and associations with health-related quality of life: results from the American Cancer Society's SCS-II. J Clin Oncol. 2008 May 1;26(13):2198-204. doi: 10.1200/JCO.2007.14.6217. PMID 18445845
- [Background] Tarasenko Y, Chen C, Schoenberg N. Self-Reported Physical Activity Levels of Older Cancer Survivors: Results from the 2014 National Health Interview Survey. J Am Geriatr Soc. 2017 Feb;65(2):e39-e44. doi: 10.1111/jgs.14589. Epub 2016 Dec 9. PMID 27943255
- [Background] Harrington JM, Schwenke DC, Epstein DR. Exercise preferences among men with prostate cancer receiving androgen-deprivation therapy. Oncol Nurs Forum. 2013 Sep;40(5):E358-67. doi: 10.1188/13.ONF.E358-E367. PMID 23989028
- [Background] Kushi LH, Doyle C, McCullough M, Rock CL, Demark-Wahnefried W, Bandera EV, Gapstur S, Patel AV, Andrews K, Gansler T; American Cancer Society 2010 Nutrition and Physical Activity Guidelines Advisory Committee. American Cancer Society Guidelines on nutrition and physical activity for cancer prevention: reducing the risk of cancer with healthy food choices and physical activity. CA Cancer J Clin. 2012 Jan-Feb;62(1):30-67. doi: 10.3322/caac.20140. PMID 22237782
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Focht BC, Lucas AR, Grainger E, Simpson C, Thomas-Ahner JM, Clinton SK. The Individualized Diet and Exercise Adherence Pilot Trial (IDEA-P) in prostate cancer patients undergoing androgen deprivation therapy: study protocol for a randomized controlled trial. Trials. 2014 Sep 9;15:354. doi: 10.1186/1745-6215-15-354. PMID 25199619
- [Background] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238
- [Background] Bourke L, Smith D, Steed L, Hooper R, Carter A, Catto J, Albertsen PC, Tombal B, Payne HA, Rosario DJ. Exercise for Men with Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Apr;69(4):693-703. doi: 10.1016/j.eururo.2015.10.047. Epub 2015 Nov 26. PMID 26632144
- [Background] Taaffe DR, Buffart LM, Newton RU, Spry N, Denham J, Joseph D, Lamb D, Chambers SK, Galvao DA. Time on androgen deprivation therapy and adaptations to exercise: secondary analysis from a 12-month randomized controlled trial in men with prostate cancer. BJU Int. 2018 Feb;121(2):194-202. doi: 10.1111/bju.14008. Epub 2017 Sep 22. PMID 28872752
- [Background] Winters-Stone KM, Dieckmann N, Maddalozzo GF, Bennett JA, Ryan CW, Beer TM. Resistance Exercise Reduces Body Fat and Insulin During Androgen-Deprivation Therapy for Prostate Cancer. Oncol Nurs Forum. 2015 Jul;42(4):348-56. doi: 10.1188/15.ONF.348-356. PMID 26148314
- [Background] Glass OK, Ramalingam S, Harrison MR. Resistance exercise training in patients with genitourinary cancers to mitigate treatment-related skeletal muscle loss. Clin Adv Hematol Oncol. 2016 Jun;14(6):436-46. PMID 27379813
- [Background] Healy GN, Dunstan DW, Salmon J, Shaw JE, Zimmet PZ, Owen N. Television time and continuous metabolic risk in physically active adults. Med Sci Sports Exerc. 2008 Apr;40(4):639-45. doi: 10.1249/MSS.0b013e3181607421. PMID 18317383
- [Background] Healy GN, Matthews CE, Dunstan DW, Winkler EA, Owen N. Sedentary time and cardio-metabolic biomarkers in US adults: NHANES 2003-06. Eur Heart J. 2011 Mar;32(5):590-7. doi: 10.1093/eurheartj/ehq451. Epub 2011 Jan 11. PMID 21224291
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Church TS, Thomas DM, Tudor-Locke C, Katzmarzyk PT, Earnest CP, Rodarte RQ, Martin CK, Blair SN, Bouchard C. Trends over 5 decades in U.S. occupation-related physical activity and their associations with obesity. PLoS One. 2011;6(5):e19657. doi: 10.1371/journal.pone.0019657. Epub 2011 May 25. PMID 21647427
- [Background] De Cocker K, Duncan MJ, Short C, van Uffelen JG, Vandelanotte C. Understanding occupational sitting: prevalence, correlates and moderating effects in Australian employees. Prev Med. 2014 Oct;67:288-94. doi: 10.1016/j.ypmed.2014.07.031. Epub 2014 Aug 10. PMID 25117522
- [Background] Lynch BM, Dunstan DW, Vallance JK, Owen N. Don't take cancer sitting down: a new survivorship research agenda. Cancer. 2013 Jun 1;119(11):1928-35. doi: 10.1002/cncr.28028. Epub 2013 Mar 15. PMID 23504979
- [Background] Benatti FB, Ried-Larsen M. The Effects of Breaking up Prolonged Sitting Time: A Review of Experimental Studies. Med Sci Sports Exerc. 2015 Oct;47(10):2053-61. doi: 10.1249/MSS.0000000000000654. PMID 26378942
- [Background] Zeigler ZS, Mullane SL, Crespo NC, Buman MP, Gaesser GA. Effects of Standing and Light-Intensity Activity on Ambulatory Blood Pressure. Med Sci Sports Exerc. 2016 Feb;48(2):175-81. doi: 10.1249/MSS.0000000000000754. PMID 26285021
- [Background] Dempsey PC, Larsen RN, Sethi P, Sacre JW, Straznicky NE, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Benefits for Type 2 Diabetes of Interrupting Prolonged Sitting With Brief Bouts of Light Walking or Simple Resistance Activities. Diabetes Care. 2016 Jun;39(6):964-72. doi: 10.2337/dc15-2336. Epub 2016 Apr 13. PMID 27208318
- [Background] Thosar SS, Bielko SL, Mather KJ, Johnston JD, Wallace JP. Effect of prolonged sitting and breaks in sitting time on endothelial function. Med Sci Sports Exerc. 2015 Apr;47(4):843-9. doi: 10.1249/MSS.0000000000000479. PMID 25137367
- [Background] Dempsey PC, Sacre JW, Larsen RN, Straznicky NE, Sethi P, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Interrupting prolonged sitting with brief bouts of light walking or simple resistance activities reduces resting blood pressure and plasma noradrenaline in type 2 diabetes. J Hypertens. 2016 Dec;34(12):2376-2382. doi: 10.1097/HJH.0000000000001101. PMID 27512975
- [Background] Gardiner PA, Eakin EG, Healy GN, Owen N. Feasibility of reducing older adults' sedentary time. Am J Prev Med. 2011 Aug;41(2):174-7. doi: 10.1016/j.amepre.2011.03.020. PMID 21767725
- [Background] Keadle SK, Conroy DE, Buman MP, Dunstan DW, Matthews CE. Targeting Reductions in Sitting Time to Increase Physical Activity and Improve Health. Med Sci Sports Exerc. 2017 Aug;49(8):1572-1582. doi: 10.1249/MSS.0000000000001257. PMID 28272267
- [Background] Bourke L, Homer KE, Thaha MA, Steed L, Rosario DJ, Robb KA, Saxton JM, Taylor SJ. Interventions to improve exercise behaviour in sedentary people living with and beyond cancer: a systematic review. Br J Cancer. 2014 Feb 18;110(4):831-41. doi: 10.1038/bjc.2013.750. Epub 2013 Dec 12. PMID 24335923
- [Background] Bourke L, Gilbert S, Hooper R, Steed LA, Joshi M, Catto JW, Saxton JM, Rosario DJ. Lifestyle changes for improving disease-specific quality of life in sedentary men on long-term androgen-deprivation therapy for advanced prostate cancer: a randomised controlled trial. Eur Urol. 2014 May;65(5):865-72. doi: 10.1016/j.eururo.2013.09.040. Epub 2013 Oct 4. PMID 24119318
- [Background] Galvao DA, Taaffe DR, Spry N, Joseph D, Newton RU. Combined resistance and aerobic exercise program reverses muscle loss in men undergoing androgen suppression therapy for prostate cancer without bone metastases: a randomized controlled trial. J Clin Oncol. 2010 Jan 10;28(2):340-7. doi: 10.1200/JCO.2009.23.2488. Epub 2009 Nov 30. PMID 19949016
- [Background] Galvao DA, Taaffe DR, Spry N, Newton RU. Exercise can prevent and even reverse adverse effects of androgen suppression treatment in men with prostate cancer. Prostate Cancer Prostatic Dis. 2007;10(4):340-6. doi: 10.1038/sj.pcan.4500975. Epub 2007 May 8. PMID 17486110
- [Background] Galvao DA, Newton RU. Review of exercise intervention studies in cancer patients. J Clin Oncol. 2005 Feb 1;23(4):899-909. doi: 10.1200/JCO.2005.06.085. PMID 15681536
- [Background] Beydoun N, Bucci JA, Chin YS, Spry N, Newton R, Galvao DA. Prospective study of exercise intervention in prostate cancer patients on androgen deprivation therapy. J Med Imaging Radiat Oncol. 2014;58(3):369-76. doi: 10.1111/1754-9485.12115. Epub 2013 Oct 4. PMID 24118798
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Trinh L, Arbour-Nicitopoulos KP, Sabiston CM, Alibhai SM, Jones JM, Berry SR, Loblaw A, Faulkner GE. A Qualitative Study Exploring the Perceptions of Sedentary Behavior in Prostate Cancer Survivors Receiving Androgen-Deprivation Therapy. Oncol Nurs Forum. 2015 Jul;42(4):398-406. doi: 10.1188/15.ONF.398-406. PMID 26148319
- [Background] Nicklas BJ, Gaukstern JE, Beavers KM, Newman JC, Leng X, Rejeski WJ. Self-monitoring of spontaneous physical activity and sedentary behavior to prevent weight regain in older adults. Obesity (Silver Spring). 2014 Jun;22(6):1406-12. doi: 10.1002/oby.20732. Epub 2014 Mar 17. PMID 24585701
- [Background] Michie S, Yardley L, West R, Patrick K, Greaves F. Developing and Evaluating Digital Interventions to Promote Behavior Change in Health and Health Care: Recommendations Resulting From an International Workshop. J Med Internet Res. 2017 Jun 29;19(6):e232. doi: 10.2196/jmir.7126. PMID 28663162
- [Background] Buman MP, Epstein DR, Gutierrez M, Herb C, Hollingshead K, Huberty JL, Hekler EB, Vega-Lopez S, Ohri-Vachaspati P, Hekler AC, Baldwin CM. BeWell24: development and process evaluation of a smartphone "app" to improve sleep, sedentary, and active behaviors in US Veterans with increased metabolic risk. Transl Behav Med. 2016 Sep;6(3):438-48. doi: 10.1007/s13142-015-0359-3. PMID 27528532
- [Background] Luger TM, Houston TK, Suls J. Older adult experience of online diagnosis: results from a scenario-based think-aloud protocol. J Med Internet Res. 2014 Jan 16;16(1):e16. doi: 10.2196/jmir.2924. PMID 24434479
- See also: Pew Internet & American Life Project. Internet/Broadband Factsheet. 2017; — http://www.pewinternet.org/fact-sheet/internet-broadband/